CLINICAL TRIAL: NCT01131156
Title: Prevention of Postpartum Smoking Relapse in Mothers of Infants in the Neonatal Intensive Care Unit
Brief Title: Prevention of Postpartum Smoking Relapse in Mothers of Infants in the Neonatal Intensive Care Unit (NICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: American Academy of Pediatrics (Other); Flight Attendant Medical Research Institute (Other); March of Dimes (Other)
Responsible Party: Principal Investigator, Raylene Phillips, MD, Medical Doctor, Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 58108
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Smoking
Keywords: postpartum; smoking; relapse; breastfeeding
MeSH Terms: conditions — Smoking; Recurrence; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Smoking Relapse Prevention — Mothers were given information about normal newborn behaviors using books, DVDs, and handouts that were appropriate for their baby's gestational age and were also encouraged to participate in frequent skin-to-skin holding of their babies.

SUMMARY:
The investigators hypothesized that an enriched focus on mother-infant bonding during a newborn's hospitalization in the Neonatal Intensive Care Unit would reduced the rate maternal postpartum smoking relapse and would prolong the duration of breastfeeding in mothers who had quit smoking during or just prior to pregnancy.

DETAILED DESCRIPTION:
Mothers of newborns admitted to the Neonatal Intensive Care Unit (NICU), who had quit smoking during or just prior to pregnancy where randomized to either the Standard of Care or Smoking Relapse Prevention group. Mothers in both groups were encouraged to remain smoke free following the birth of their babies and were given routine lactation support for breastfeeding during their babies' hospitalization in the NICU. Mothers in the Smoking Relapse Prevention group were also given the study intervention, which was enhanced support for maternal-infant bonding by providing information about their newborn's behaviors using books, DVDs, and handouts that were appropriate for their baby's gestational age and by encouraging frequent skin-to-skin holding.

Primary outcomes included duration of smoke-free status and duration of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Mothers:

  * Who had quit smoking during pregnancy or within one year prior to pregnancy
  * Who had newborns < 1 week old at the time of admission to our NICU.

Exclusion Criteria:

* Mothers:

  * Who were smokers at the time of delivery
  * Whose infant's length of stay < one week
  * Who were not available (jail, adoption)
  * Who had a history of drug use
  * Who did not speak English

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Duration of smoke-free status | 8 weeks postpartum
  Duration of maternal smoke-free status during the first 8 weeks postpartum following delivery of newborn infant
Duration of breastfeeding | 8 weeks postpartum
  Duration of breastfeeding during the first 8 weeks postpartum following the birth of newborn infant.

CONTACTS AND LOCATIONS:
Overall Officials: T. Allen Merritt, MD, MHA, Principal Investigator — Loma Linda University, School of Medicine
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States